CLINICAL TRIAL: NCT00511745
Title: Safety of Rabeprazole in Patients Under Multiple Treatments
Status: Terminated | Type: Observational
Why Stopped: Due to the achievement of minimum required sample size and new changes in local regulations.
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR009238
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux; Gastric Ulcer
Keywords: Interactions; Adjusted doses; Duodenal Ulcer; Gastric Ulcer; Erosive or ulcerate Gastroesophageal Reflux; Rabeprazole; Gastroesophageal reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Stomach Ulcer; Duodenal Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Rabeprazol

INTERVENTIONS:
Drug: Rabeprazol — As prescribed

SUMMARY:
The purpose of this study is to evaluate the safety of rabeprazole 20mg/day in polymedicated patients and to examine the necessity of adjusted dosage in both therapies (rabeprazole and concomitant drug). Proton pump inhibitors (PPI) act in the final step of the gastric secretion. PPI's block ATP-ase H+/K+ in gastric parietals cells. It has been described that inhibition of acid secretion has produced the recovery of the gastroesophageal pathology in a high percentage of the patients resistant to conventional drugs. In this context, the objective of the study is to evaluate the safety of rabeprazole as a concomitant treatment and examine the clinical practice the interaction with drugs whose absorption has gastric pH dependence.

DETAILED DESCRIPTION:
Rabeprazole is a new proton pump inhibitor (PPI) with potent anti-secretion action and dose-dependence activity. Rabeprazole is rapidly eliminated by hepatic metabolism and renal clearance. In previous studies in healthy volunteers, interactions between sodium rabeprazole and drugs such as warfarin, theophyline, diazepam and phenytoin have not been found. The objective of the study is to evaluate the safety of rabeprazole as concomitant treatment and examine the clinical practice of the interaction with drugs whose absorption has a gastric pH dependence. This is an observational, multicenter, open and prospective study. It is expected to enroll 500 patients receiving rabeprazole and a concomitant drug (one or more). All data collected will be prospective and will include the following: demographic data, adherence and compliance with treatment, lifestyle (smoking and alcohol consumption) and dose of rabeprazole. Safety analysis will be based on adverse events. Observational Study: For patients with duodenal or gastric ulcer: rabeprazole 20mg per day, orally, for 4-6 weeks; For patients with erosive or ulcerate gastroesophagic reflux: rabeprazole orally 20mg/ per day, 4-8 weeks; For patients with gastroesophagic reflux requiring prolonged treatment: rabeprazole orally 10 or 20 mg per day; For patients with H. Pylori: rabeprazole orally 20mg twice per day , Clarithromycin orally 500mg 2 times per day and Amoxicillin 1gram orally twice daily for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Rabeprazole and a concomitant drug (one or more) such a non-steroidal anti-inflammatory drugs (NSAID), benzodiazepines or corticoids

Exclusion Criteria:

* Pregnant or lactating patients
* Other severe concomitant pathologies
* History or drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving rabeprazole and a concomitant drug (one or more) such a non-steroidal anti-inflammatory drugs (NSAID), benzodiazepines or corticoids
Sampling Method: Non-Probability Sample
Enrollment: 2157 (Actual)
Dates: Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Safety of rabeprazole 20mg/day in polymedicated patients | 2 or 8 weeks, as per investigator criteria

SECONDARY OUTCOMES:
No secondary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Safety of rabeprazole in patients under multiple treatments. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=282&filename=CR009238_CSR.pdf